CLINICAL TRIAL: NCT01538186
Title: Treatment Of Coronary Bifurcation Lesions: Stentcovering Of The Side Branch With And Without PCI Of The Side Branch: A Retrospective Analysis Of All Consecutive Patients
Status: Completed | Type: Observational
Sponsor: Krankenhaus Hetzelstift (Other)
Responsible Party: Principal Investigator, Hubertus von Korn, MD, Head of the Department, Krankenhaus Hetzelstift
Other Study IDs: Hetzel01
Record Dates: First submitted 2012-02-17; First posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Bifurcation Lesions
Keywords: Coronary intervention; PCI of the side branch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCI without treating the side branch
- PCI with treating the side branch

SUMMARY:
This retrospective observational study included patients (pts) with percutaneous coronary intervention (PCI) of a de novo coronary bifurcation lesion in one German center between January 2008 - August 2011. The investigators included all consecutive patients where the side branch was covered with a stent. Patients with ACS/cardiogenic shock were not excluded.

Two different methods were compared: group A represents patients with a simple strategy without any treatment of the side branch (SB). Group B consisted of patients where the SB was treated (PCI and/or stenting).

For the treatment of bifurcation lesions we used the concept of "provisional stenting", indications for the treatment of the SB were residual stenosis > 50 %, TIMI flow reduction < 2. Final-kissing PCI was intended in all patients of group B.

MACE during follow-up was evaluated in all patients.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with a bifurcation lesion, where the side branch was covered with a stent placed inside the main branch.

Exclusion Criteria:

* Patients with an in-stent-restenosis, patients with a therapy using a drug coated balloon during the procedure (inside the main branch and/or the side branch) and patients where the side branch was not covered by the stent inside the main branch.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective observational study included patients (pts) with PCI of a de novo coronary bifurcation lesion in one German center between January 2008 - August 2011. We included all consecutive patients where the side branch was covered with a stent. Patients with ACS/cardiogenic shock were not excluded.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac outcome | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hetzelstift, Neustadt/Weinstrasse, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] von Korn H, Stefan V, van Ewijk R, Chakraborty K, Sanwald B, Andel R, Hemker J, Hink U, Ohlow M, Lauer B, Muenzel T. Treatment of coronary bifurcation lesions: stent-covering of the side branch with and without PCI of the side branch: a retrospective analysis of all consecutive patients. BMC Cardiovasc Disord. 2013 Apr 4;13:27. doi: 10.1186/1471-2261-13-27. PMID 23557395